CLINICAL TRIAL: NCT01633346
Title: Regulation of the Immune System in Response to the Treatment With Tocilizumab in RA Patients
Brief Title: Regulation of the Immune System in Response to the Treatment With Tocilizumab in Rheumatoid Arthritis Patients
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: KUL-TOC-2010-01
Record Dates: First submitted 2012-06-28; First posted 2012-07-04 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tocilizumab treated patients: Rheumatoid arthritis patients

SUMMARY:
The purpose of this study is to know the level of expression and activation state of different transcription factors of the STAT family (STAT1, STAT3, STAT5A, STAT5B, STAT6) in the hematopoietic cells from tocilizumab treated patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe active RA of ≥6 months duration.
* Patients who have commenced treatment with Ro-Actemra® (tocilizumab) in accordance with the approved Summary of Product Characteristics.
* Age > 18 years.
* Body weight ≤150 kg.
* Non-pregnant, non-nursing female, and females of child-bearing potential must use a reliable means of contraception, eg, physical barrier (patient and partner), contraceptive pill or patch, spermicide and barrier, or intrauterine device (IUD)
* If female and of childbearing potential, the patient must have a negative urine at screening and baseline.
* If patients are receiving an oral corticosteroid, the prednisone dose or its equivalent must be ≤10 mg/day and stable for ≥28 days prior to screening.
* If patients are currently taking a permitted non-biologic DMARD, the dose must be stable for ≥7 weeks prior to baseline. Willing to receive oral folate or leucovorin if taking methotrexate.
* Patients who have been given written information about the study and have consented to data collection and review.

Exclusion Criteria:

* History of autoimmune disease or inflammatory joint disease other than RA.
* Treatment with any investigational agent within 4 weeks (or 5 half-lives of investigational agent, whichever is longer) before starting treatment with Ro-Actemra®
* Pregnant women or nursing (breastfeeding) mothers
* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following randomization.
* Functional class IV as defined by the ACR Classification of Functional Status in RA (ie, largely or wholly incapacitated with patient bedridden or confined to wheel chair, permitting little or no self-care)
* Treatment with rituximab within 6 months before screening.
* Treatment with IV gamma globulin, plasmapheresis or Prosorba® column within months, or any investigational cell-depleting therapies before baseline.
* Immunization with a live/attenuated vaccine within 4 weeks prior to baseline.
* Any previous treatment with alkylating agents, such as cyclophosphamide or chlorambucil, or with total lymphoid irradiation.
* Treatment with:

Intraarticular (IA) corticosteroids within 8 weeks prior to screening. Intramuscular (IM) or IV corticosteroids within 12 weeks prior to screening.

* History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies.
* Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine(including uncontrolled diabetes mellitus) or GI disease (including complicated
* Evidence of active malignant disease, malignancies diagnosed within the previous 5 years (including hematological malignancies and solid tumors, except non melanoma skin cancer that has been excised and cured), or breast cancer diagnosed within the previous 5 years.
* Active TB requiring treatment within the previous 3 years. Patients previously treated for TB with no recurrence in the past 3 years are permitted. Patients who have a positive purified protein derivative (PPD) tuberculin skin test and have not been adequately treated for TB must be treated for latent TB with isoniazid (INH) for 1 month prior to enrollment whether or not they have been vaccinated in the past. Patients with a positive PPD that is ≥5mm at screening are not eligible for the study unless they begin treatment for latent TB with INH a minimum of 1 month prior to enrollment in the trial. The required total INH treatment duration is 9 months. Patients must have a negative CXR at enrollment.
* HIV-positive.
* History of alcohol, drug or chemical abuse within the 6 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with RA who are going to commence treatment with Ro-Actemra® (Tocilizumab). All patients initiating treatment will be considered for the study if they fulfill all inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-06; Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Changes in the levels of phosphorylation of STAT proteins on peripheral blood leukocytes | 6 months
  The levels of phosphorylation of STATs on different subsets of leukocytes will be assessed by flow cytometry at baseline (before Tocilizumab administration) and at the indicated time (6m) after initiation of treatment. Results will be expressed as Mean of Fluorescence Intensity. To perform the analysis the investigators will use conjugated monoclonal antibodies against STAT1, STAT3, STAT5 and STAT6

SECONDARY OUTCOMES:
Main change in plasma level of IL-2, IL-4, IL-6, IL-10, IL-17, TNFα, IFNα, IFNγ,MCP-1 and IL-1 | Baseline, at month 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Vidal, PhD, Principal Investigator — Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain